CLINICAL TRIAL: NCT00008177
Title: A Phase I Study Combining Escalating Doses of Radiolabeled BC8 (Anti-CD45) Antibody With Fludarabine, Low Dose TBI, PBSC Infusion and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil to Establish Mixed or Full Donor Chimerism for Elderly Patients With Advanced Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Brief Title: Radiolabeled Monoclonal Antibody Therapy, Fludarabine Phosphate, and Low-Dose Total-Body Irradiation Followed by Donor Stem Cell Transplant and Immunosuppression Therapy in Treating Older Patients With Advanced Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1432.00; NCI-2010-02046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1432; 1432.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA044991 (NIH)
Record Dates: First submitted 2001-01-06; First posted 2003-12-12 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; fludarabine phosphate; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment ( I 131 BC8, chemotherapy, TBI, PBSCT, CSP, MMF) (Experimental): CONDITIONING REGIMEN: Patients receive iodine I 131 monoclonal antibody BC8 IV on day -12 and fludarabine phosphate IV on days -4 to -2. Patients undergo total-body irradiation on day 0.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO or IV BID on days -3 to 56 with taper to day 80 (for patients with a related donor) OR days -3 to 100 with taper to day 177 (for patients with an unrelated donor) in the absence of GVHD. Patients also receive mycophenolate mofetil PO or IV TID on days 0 to 27 (for patients with a related donor) OR on days 0 to 40 with taper to day 96 (for patients with an unrelated donor) in the absence of GVHD.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: fludarabine phosphate; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody BC8 — Given IV
  Other Names: I 131 MOAB BC8; I 131 Monoclonal Antibody BC8; iodine I 131 MOAB BC8
Radiation: total-body irradiation — Undergo total-body irradiation
  Other Names: TBI
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplantation
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclosporine — Given orally or IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given orally or IV
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of iodine I 131 monoclonal antibody BC8 when given together with fludarabine phosphate and low-dose total-body irradiation followed by donor stem cell transplant and immunosuppression therapy in treating older patients with acute myeloid leukemia or high-risk myelodysplastic syndromes that cannot be controlled with treatment. Radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them. Giving chemotherapy, such as fludarabine phosphate, and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer or abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving radiolabeled monoclonal antibody therapy together with fludarabine phosphate and total-body irradiation before the transplant together with cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of radiation delivered via 131I-BC8 antibody (iodine I 131 monoclonal antibody BC8) when combined with the non-myeloablative regimen of fludarabine (fludarabine phosphate), 2 Gy total-body irradiation (TBI) + cyclosporine (CSP)/mycophenolate (MMF) in elderly patients with advanced acute myeloid leukemia (AML) or high risk myelodysplastic syndromes (MDS).

II. To determine the rates of donor chimerism resulting from this combined preparative regimen, and to correlate level of donor chimerism with estimated radiation doses delivered to hematopoietic tissues via antibody.

III. To determine, within the limits of a phase I study, disease response and duration of remission.

IV. To assess dose-limiting toxicity (DLT) at the estimated maximum tolerated dose (MTD) of 131I-BC8 (24 Gy) in order to gain more confidence that the DLT rate is acceptable at this level.

OUTLINE: This is a dose-escalation study of iodine I 131 monoclonal antibody BC8.

CONDITIONING REGIMEN: Patients receive iodine I 131 monoclonal antibody BC8 intravenously (IV) on day -12 and fludarabine phosphate IV on days -4 to -2. Patients undergo total-body irradiation on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) or IV twice daily (BID) on days -3 to 56 with taper to day 80 (for patients with a related donor) OR days -3 to 100 with taper to day 177 (for patients with an unrelated donor) in the absence of graft-versus-host disease (GVHD). Patients also receive mycophenolate mofetil PO or IV thrice daily (TID) on days 0 to 27 (for patients with a related donor) OR on days 0 to 40 with taper to day 96 (for patients with an unrelated donor) in the absence of GVHD.

After completion of study treatment, patients are followed up at 6, 9, and 12 months, every 6 months for 1 year, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced AML defined as beyond first remission, primary refractory disease, or evolved from myelodysplastic or myeloproliferative syndromes; or patients with MDS expressed as refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEBT [Note: classification removed under current World Health Organization [WHO] classification system]), refractory cytopenia with multilineage dysplasia (RCMD), RCMD with ringed sideroblasts (RCMD-RS), or chronic myelomonocytic leukemia (CMML)
* Patients in relapse must have documented cluster of differentiation (CD)45 expression by their myelodysplastic or leukemic cells to be studied and treated with 131I-labeled BC8 antibody; patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed)
* Patients must undergo a 24-hour urine collection with documented creatinine clearance > 50 ml/min
* Bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times the upper limit of normal
* Karnofsky score >= 70 or Eastern Cooperative Oncology Group (ECOG) =< 2
* Patients must have an expected survival of > 60 days and must be free of active infection
* Patients must have a human leukocyte antigen (HLA)-identical sibling donor or an HLA-matched unrelated donor who meets standard Seattle Cancer Care Alliance (SCCA) and/or National Marrow Donor Program (NMDP) criteria for peripheral blood stem cell (PBSC) donation; related donors should be matched by molecular methods at the intermediate resolution level at HLA-A, B, C, and DRB1 according to Fred Hutchinson Cancer Research Center (FHCRC) Standard Practice Guidelines and to the allele level at DQB1; unrelated donors should be identified using matching criteria that follows the FHCRC Standard Practice Guidelines limiting the study to eligible donors that are allele matched for HLA-A, B, C, DRB1, and DQB1 (grade 1), and accepting up to one allele mismatch as per standard practice grade 2.1 for HLA-A, B, or C; PBSC is the only permitted hematopoietic stem cell (HSC) source
* DONOR: Donors must meet HLA matching criteria as outlined above as well as standard Seattle Cancer Care Alliance (SCCA) and/or NMDP criteria for PBSC donation

Exclusion Criteria:

* Circulating antibody against mouse immunoglobulin (human anti-mouse antibody [HAMA])
* Prior radiation to maximally tolerated levels to any normal organ
* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects
* Inability to understand or give an informed consent
* Patients who are seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures, particularly treatment in radiation isolation
* Patients who have previously undergone marrow or PBSC transplantation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 1999-07-27 (Actual); Primary Completion 2009-03-21 (Actual); Study Completion 2010-12-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of radiation delivered via 131I-BC8 antibody when combined with the nonmyeloablative regimen of fludarabine phosphate, TBI, and CSP/MMF | Up to day 100 following transplant
Rates of donor chimerism resulting from this combined preparative regimen | Up to day 84 following transplant
  Correlated with estimated radiation doses delivered to hematopoietic tissues via antibody.
Disease response | Up to 11 years
Duration of remission | Up to 11 years
incidence of DLT at the estimated MTD of 131I-BC8 | Up to day 100 following transplant

CONTACTS AND LOCATIONS:
Overall Officials: Johnnie Orozco, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Pagel JM, Gooley TA, Rajendran J, Fisher DR, Wilson WA, Sandmaier BM, Matthews DC, Deeg HJ, Gopal AK, Martin PJ, Storb RF, Press OW, Appelbaum FR. Allogeneic hematopoietic cell transplantation after conditioning with 131I-anti-CD45 antibody plus fludarabine and low-dose total body irradiation for elderly patients with advanced acute myeloid leukemia or high-risk myelodysplastic syndrome. Blood. 2009 Dec 24;114(27):5444-53. doi: 10.1182/blood-2009-03-213298. Epub 2009 Sep 28. PMID 19786617